CLINICAL TRIAL: NCT02534714
Title: Analysis of Hypovitaminosis D and Osteopenia/Osteoporosis in Spinal Disease Patients Who Underwent a Spinal Fusion at Illinois Neurological Institute, Peoria, IL., a Retrospective Review From November 1, 2012 to October 31, 2014 and Prospective Pilot From July 1, 2015-June 30, 2016
Status: Completed | Type: Observational
Sponsor: OSF Healthcare System (Other)
Collaborators: University of Illinois College of Medicine at Peoria (Other)
Responsible Party: Principal Investigator, Jana Reed, Jana Reed, APN, OSF Healthcare System
Other Study IDs: 632002
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Hypovitaminosis D; Spinal Disease; Osteoporosis
MeSH Terms: conditions — Vitamin D Deficiency; Spinal Diseases; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective (Part 1) Group: This is a retrospective pilot study in patients diagnosed with any form of spinal disease who underwent spinal fusion at OSF/INI by Dr. Daniel Fassett, MD, MBA, Neurosurgeon from November 1, 2012 to October 31, 2014. Only spinal fusion patients with a serum Vitamin D level prior to or at time of surgery and after surgery are included in this review. The following variables will be utilized to characterize the sample: age, sex, ethnicity, BMI, smoking history, pre-op Vitamin D level and supplement given. The charts reviewed will belong to subjects who were closely followed at the OSF/INI clinic.
- Prospective (Part 2) Group: This is a prospective pilot study in subjects diagnosed with any form of spinal disease that underwent cervical, thoracic, and/or lumbar spinal fusion at OSF/INI by Dr. Daniel Fassett, MD, MBA, Neurosurgeon from July 1, 2015 to June 30, 2016.
  (Screening period July 1, 2015-June 30, 2016)
  Only spinal fusion patients with a serum Vitamin D level, and Bone Marrow Density prior to or at time of surgery are included in this study. The following variables will be utilized to characterize the sample: age, sex, ethnicity, BMI, smoking history, pre-op Vitamin D level and supplement given. The subjects were closely followed at the OSF/INI clinic post-operatively at 3, 6, and 12 months. Pre-op Vitamin D level and Bone Marrow Density will be measured at the baseline, and again at 3, 6, and 12 months.

SUMMARY:
The purpose of this study is to determine if there is correlation between Vitamin D deficiency and spinal disease/spinal fusion surgery.

DETAILED DESCRIPTION:
Bone Health is becoming of great concern in the population > 50 years old in the past several decades. Literature review has detected a high incidence of patients with hypovitaminosis D and back pain. Vitamin D Deficiency is in all races, age groups, and ethnic backgrounds affecting greater than one billion people worldwide1. There is a higher incidence of Vitamin D Deficiency noted in the northern states.

Adequate Vitamin D is essential in bone health and muscle function. It also has been reported to have positive effects on decreasing myopathy and /or musculoskeletal pain. Vitamin D has been shown to have a protective effect on fracture risk by providing increased bone matrix and on fall prevention through improved muscle function. 2

Deficiency of this vitamin can lead to impaired bone mineralization and bone softening diseases including osteomalacia and osteoporosis in adults. Osteomalacia has significant risk factors for vertebral fractures, and spinal instrumentation failure. Low-energy fractures or fragility fractures have been found to be more common because of an increase in life expectancy 3. The total 25-hydroxyvitamin D (25-OH-VitD) level (the sum of 25-OH-vitamin D2 and 25-OH-vitamin D3) is the appropriate indicator of vitamin D body stores. Presently, there is no universal consensus about a treatment cut point. Studies suggest >30 ng/mL as the minimal concentration of 25-OH-Vit D Total is needed to avoid the adverse effects of deficiency4. Vitamin D insufficiency is considered at <30ng/ml to 21 ng/ml and Vitamin D Deficiency is <20 ng/ml of 25-OH-Vit D Total. Several researches have indicated increasing Vitamin D levels >45 ng/ml will increase their immune system, bone health, lower risks of neurological disorders and cancers. 3,4

Influential pathophysiological changes in osteoporosis include the hyperactivity of osteoclasts compared to the need for bone remodeling or a decreased activity of osteoblasts compared to the need for bone cavity repair or laying down new bone.5 Osteoporosis has become synonymous with decreased bone mineral density (BMD). Bone Marrow Density scans (DXA) allows accurate diagnosis of osteoporosis, estimation of fracture risk, and monitoring of patients undergoing treatment.5 In postmenopausal women and men age 50 years and older, the WHO diagnostic T-score criteria categorizes a normal DXA scan of <1.0 or above, low bone mass or osteopenia has a T score between <1.0 and -2.5, and osteoporosis is designated with a T-score at -2.5 or below) are applied to BMD measurement by central DXA at the lumbar spine and femoral neck. 5

This study was done in two parts. Part 1 was the Retrospective Study from November 1, 2012 to October 31, 2014 and Part 2 is the Prospective pilot from July 1, 2015-June 30, 2016. We are anticipating to raise the awareness and identify the importance of evaluating for hypovitaminosis D and bone marrow density preoperatively in Neurosurgery Clinic for 12 months. Our goal is to show treating bone health in spinal diseased patients preoperatively will provide optimal bone health with better long term outcomes requiring less revision surgeries for our patients.

Research Question:

Part 1 - Retrospective Study

1. What is the prevalence of Vitamin D Deficiency in patients over 50 undergoing spinal fusion surgery by Dr. Daniel Fassett, MD, MBA, Neurosurgeon?

Part 2- Prospective Study (screening period July 1, 2015-June 30, 2016)

1. What is the prevalence of Vitamin D Deficiency in patients over 50 undergoing spinal fusion surgery by Dr. Daniel Fassett, MD, MBA, Neurosurgeon?
2. Do patients with Hypovitaminosis D maintain therapeutic levels between 45 ng/ml to 75 ng/ml in approximately 3, 6, and 12 months postoperatively with supplements of Vitamin D3?
3. What are the incidences of osteopenia and osteoporosis in elective spinal fusion patients based on a Dexascans in patients over 50 undergoing spinal fusion surgery by Dr. Daniel Fassett, MD, MBA, Neurosurgeon?
4. Do the patients' demographic information, such as age, sex, BMI, and family history influence the outcome measures (Vitamin D deficiency, Osteopenia, and Osteoporosis)?

ELIGIBILITY:
(Part 1, Retrospective Study)

Inclusion Criteria:

1. 50 years old or older.
2. Patients with any form of spinal fusion surgery performed by Dr. Daniel Fassett, MD, MBA, Neurosurgeon at OSF-INI from November 1, 2012 to October 31, 2014.

   Exclusion Criteria:
3. Subjects diagnosed with chronic renal disease Stage IV or V, metastatic spinal disease, bariatric surgery, malabsorption syndrome, seizure medication and chronic steroid use greater than 3 months at time of surgery.

(Part 2, Observational Study)

(Screening period July 1, 2015-June 30, 2016)

Inclusion Criteria:

1. 50 years old or older.
2. Serum Vitamin D level checked prior to or at surgery.
3. BMD exam performed anytime within 2 years prior to surgery.
4. Patients with any form of spinal fusion cervical, thoracic, lumbar, surgery performed by Dr. Daniel Fassett, MD, MBA, Neurosurgeon at OSF-INI from July 1, 2015 to May 31, 2016.

   Exclusion Criteria:
5. Subjects diagnosed with:

   * Chronic Renal Disease with a GFR < 45 at Stage IV
   * Metastatic Spinal Disease
   * Bariatric surgery
   * Seizure medication
   * Chronic steroid use greater than 3 months at time of surgery.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (Part 1, Retrospective Study) - patients diagnosed with any form of spinal disease who underwent spinal fusion at OSF/INI by Dr. Daniel Fassett, MD, MBA, Neurosurgeon from November 1, 2012 to October 31, 2014 who had a serum vitamin D level collected as standard of care prior to surgery.
  (Part 2, Prospective Study) - patients diagnosed with any form of spinal disease that underwent cervical, thoracic, and/or lumbar spinal fusion at OSF/INI by Dr. Daniel Fassett, MD, MBA, Neurosurgeon from July 1, 2015 to June 30, 2016 who had a serum vitamin D level and bone marrow density scan collected as standard of care prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
(Part 1, Retrospective Study) Serum vitamin D 25 Hydroxy Level | Within 30 days (pre-op)
  Prospective Vitamin D lab of 25 Hydroxyvitamin D Total <30 ng/ml in the population >50 years old will have increased incidence of progressive spinal disease.
(Part 2, Prospective Study) Serum vitamin D 25 Hydroxy Level | Pre-op and at 3, 6, 12 months post-op
  1. Vitamin D values. We will categorize it to different levels: if the value is <30 ng/ml to 21 ng/ml-then it is insufficient; if the value is <20 ng/ml, then it is deficient.
(Part 2, Prospective Study) Bone Marrow Density Results (DMD, DEXA) | Within 2 years prior to spinal surgery
  Categorized as normal, osteopenia, and osteoporosis

SECONDARY OUTCOMES:
(Part 1) Demographics | Screening
  Gender, Age, Ethnicity
(Part 1) Medical History | Screening - immediately post-op
  Medical History, BMI, smoking status, supplementation
(Part 2) Demographics | Screening
  Gender, Age, Ethnicity
(Part 2 ) Medical History | Screening - 12 months post-op
  Family history osteoporosis, smoking status, calcium and vitamin D supplementation, and diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Todd McCall, MD, Study Chair — OSF Saint Francis, Illinois Neurological Institute; Jana Reed, APN, Principal Investigator — OSF Saint Francis Medical Center, Illinois Neurological Institute
Locations (1):
- OSF Saint Francis Medical Center, Peoria, Illinois, United States

REFERENCES:
- [Background] Bogunovic L, Kim AD, Beamer BS, Nguyen J, Lane JM. Hypovitaminosis D in patients scheduled to undergo orthopaedic surgery: a single-center analysis. J Bone Joint Surg Am. 2010 Oct 6;92(13):2300-4. doi: 10.2106/JBJS.I.01231. PMID 20926724
- [Background] Kim TH, Yoon JY, Lee BH, Jung HS, Park MS, Park JO, Moon ES, Kim HS, Lee HM, Moon SH. Changes in vitamin D status after surgery in female patients with lumbar spinal stenosis and its clinical significance. Spine (Phila Pa 1976). 2012 Oct 1;37(21):E1326-30. doi: 10.1097/BRS.0b013e318268ff05. PMID 22805343
- [Background] Dipaola CP, Bible JE, Biswas D, Dipaola M, Grauer JN, Rechtine GR. Survey of spine surgeons on attitudes regarding osteoporosis and osteomalacia screening and treatment for fractures, fusion surgery, and pseudoarthrosis. Spine J. 2009 Jul;9(7):537-44. doi: 10.1016/j.spinee.2009.02.005. Epub 2009 Mar 28. PMID 19328744
- [Background] Heaney RP. Vitamin D: how much do we need, and how much is too much? Osteoporos Int. 2000;11(7):553-5. doi: 10.1007/s001980070074. No abstract available. PMID 11069187
- [Background] Manolagas SC. Birth and death of bone cells: basic regulatory mechanisms and implications for the pathogenesis and treatment of osteoporosis. Endocr Rev. 2000 Apr;21(2):115-37. doi: 10.1210/edrv.21.2.0395. PMID 10782361
- [Background] Blake GM, Fogelman I. The role of DXA bone density scans in the diagnosis and treatment of osteoporosis. Postgrad Med J. 2007 Aug;83(982):509-17. doi: 10.1136/pgmj.2007.057505. PMID 17675543